CLINICAL TRIAL: NCT04065256
Title: Effects of Music Therapy on Reducing Delirium in Mechanically Ventilated Adults in Intensive Care Unit: a Randomized Controlled Trial
Brief Title: Effects of Music Therapy on Reducing Delirium in Mechanically Ventilated Adults in Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Associated professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N201905008
Record Dates: First submitted 2019-08-16; First posted 2019-08-22 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Critical Illness; Mechanical Ventilation
Keywords: music therapy; intensive care unit; delirium
MeSH Terms: conditions — Critical Illness; Delirium | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized music intervention group (Experimental): Participants will receive a personalized music session for forty minutes twice a day for consecutive seven days or until discharge from ICU. A total treatment dosage of 560 minutes is required.
  Interventions: Other: Personalized music
- Personalized music plus earplug group (Experimental): Participants will receive a personalized music session for forty minutes twice a day for consecutive seven days or until discharge from ICU. In addition, using earplug during night time sleep. The music intervention total treatment dosage of 560 minutes is required.
  Interventions: Other: Personalized music plus earplug
- Control group (No Intervention): The control group involves neither music intervention nor using earplug at night.

INTERVENTIONS:
Other: Personalized music — Personalized music intervention will be conducted by research nurse independently. Firstly, the music preference will be confirmed by using predesigned music list. After confirming the music preference, participants will receive a music session for forty minutes through headphone and MP3 player.
  Arms: Personalized music intervention group
Other: Personalized music plus earplug — Personalized music intervention will be conducted by research nurse independently. Firstly, the music preference will be confirmed by using predesigned music list. After confirming the music preference, participants will receive a music session for forty minutes through headphone and MP3 player. In addition, participants will be worn earplug during night time sleep for decreasing the noise until next morning.
  Arms: Personalized music plus earplug group

SUMMARY:
Background: Delirium is a common acute confusion state in patients in intensive care units (ICUs). It has been linked to poor clinical prognoses (e.g., prolonged ICU stay) in critical patients. Furthermore, it might connect with long-term cognitive dysfunction. Mostly, pharmacological treatments have been frequently prescribed for preventing ICU delirium; however, their side effects might subsequently increase the risks of ICU delirium. Therefore, developing an effective non-pharmacological intervention of preventing delirium among critically mechanical ventilated patients is of clinical relevance. Purposes: To examine the effects of music intervention on reducing delirium in mechanically ventilated critical patients, to determine its beneficial effects on delirium-related outcomes, including sedation time, the duration of mechanical ventilation, and the length of ICU stay, and to compare the change of heart rate variability between groups.

DETAILED DESCRIPTION:
Delirium is a common acute confusion state among critical patients in intensive care units (ICUs). The symptoms are serious disturbance in mental abilities which may cause inattention, confused thinking, agitated mood, and fluctuated consciousness. Delirium also lead to higher mortality, longer hospital stay, higher cost of healthcare and poor recovery. However, the mechanism of delirium still not fully understand. Imbalanced neurotransmitters may be one of the possible explain for such situation. It is related to increased level of dopamine and acetylcholine deficiency. In addition, the relation between low level of melatonin and postoperative delirium was also reported. Glucocorticoid which represent the stress response is also related to postoperative delirium. Both changes of neurotransmitters and hormone levels would affect sleep-awake cycle. It is observed that patients who is delirium show a relative higher EEG theta power and a reduced alpha power than non-delirious patients. Several modifiable risk factors, such as noise, light, physical restrain, pain, anxiety, and sedatives, may contribute to poor sleep quality or sleep disruption and further delirium occurrence. Effectiveness interventions are extremely important when patients are inevitably exposed to such risk factors.

Pharmacological interventions are rapid and effective way for delirium management. However, the concern about side effect and increased mortality among high risk patients are needed. According to 2018 Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU, non-pharmacological intervention was suggested for delirium management firstly. Non-pharmacological interventions, such as using earplug or eye mask at night, music therapy or early mobilization, should be safe, less side effect and widely applicable for first-line healthcare providers. In addition, multicomponent interventions should be more effective than single component intervention. However, the evidence of direct comparison is limited.

Music intervention is a non-invasive, low-cost and non-pharmacological intervention. Several clinical trials were proved that music therapy could reduce the pain and anxiety among postoperative and old age population for better clinical progress. Listening to soft music can enhance brain alpha wave, and there is a negative correlation between alpha wave of EEG and sympathetic excitation. The preference of music also influences power of alpha wave. Recent studies report that implying music intervention on postoperative patients could lead to fewer acute confusion status, however, the incidence and potential exposed risk factors of delirium between medical and surgical populations were different. The effect of music intervention on medical critical patients and the related mechanism still need further investigation. In addition, whether the multicomponent intervention could obtain greater effect than single component intervention still not ascertained. Furthermore, the evidences of music intervention in decreasing the duration of mechanical ventilation, length of ICU stay, sedation time and mortality were still lacking. The mechanism between music intervention and delirium occurrence also need to further investigate.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 20 to 85 years
2. Expected to receive mechanical ventilation more than 24 hours
3. Be able to communicate with others using verbal or non-verbal (such as paper and pencil) approaches when enrollment.

Exclusion Criteria:

1. Dementia
2. Psychiatric illness
3. Suspected or confirmed drug or alcohol intoxication/overdose or withdrawal
4. Severe or uncorrected hearing impairment
5. Coma status after cardiac arrest or/and hypothermia treatment
6. Deep sedation needed (RASS=-4~-5 or SAS=1~2)
7. Expected death within 24h
8. Delirium history during this admission
9. Attending physician or healthcare team refusal

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Delirium incidence | Date of study enrollment through 7th day, or date of discharge from ICU.
  The number of patients who with delirium. The delirium event is assessed by Intensive Care Delirium Screening Checklist (ICDSC).
Delirium/ coma free days | Date of study enrollment through 7th day, or date of discharge from ICU.
  The number of days that free from delirium or coma status

SECONDARY OUTCOMES:
Sedation level | Date of study enrollment through 7th day, or date of discharge from ICU.
  Sedation level is assessed by Richmond Agitation-Sedation Scale (RASS). It is a ranking scale with 10-level (+4 "combative" to -5 "unarousable") used to measure the agitation or sedation level of a person. RASS score will be reported.
Pain score | Date of study enrollment through 7th day, or date of discharge from ICU.
  Pain score is assessed by Critical-Care Pain Observation Tool (CPOT). CPOT score will be reported.
Sleep quality | Date of study enrollment through 7th day, or date of discharge from ICU.
  Sleep parameters are measured by mini motionlogger actigraph. Sleep parameters will be reported.
Change from baseline on heart rate variability (HRV) | The date of enrollment, the 4th day, and the 7th day.
  Heart rate variability is measured by portable ECG recorder and analyzer.
Duration of mechanical ventilation | Date of study enrollment through weaning from mechanical ventilation, or date of study enrollment up to 90 days.
  The total days of mechanical ventilation.
Length of ICU stay | Date of study enrollment through discharge from ICU, or date of study enrollment up to 90 days.
  The total days of ICU stay.
Sedation time | Date of study enrollment through 7th day or discharge from ICU
  The total time of sedation drug used.
Mortality | The time points of measurement are 30th and 90th days.
  The number of death in a period of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, Taipei, Taiwan